CLINICAL TRIAL: NCT06683716
Title: Remote Assistance Via Smart Glasses Compared to In-person Assistance for Cannulation of the Native Papilla During Endoscopic Retrograde Cholangiopancreatography
Brief Title: SmartGlass-Guided ERCP with Cannulation of Native Papilla 1.0
Acronym: EmeRald
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Kliniken Schwerin (Other)
Responsible Party: Principal Investigator, Dr. med. Daniel Schmitz, Head physician of the Department of Gastroenterology, Helios Kliniken Schwerin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Helios SN GAS 2024-11-01
Record Dates: First submitted 2024-11-01; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Biliary Tract Diseases; Pancreatic Diseases
Keywords: Telemedicine; Training Technique; Cholangiopancreatography, Endoscopic Retrograde
MeSH Terms: conditions — Biliary Tract Diseases; Pancreatic Diseases

STUDY DESIGN:
Intervention Model Description: Prospective randomised non-inferiority trial comparing two training conditions in gastrointestinal endoscopy (ERCP)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training in presence (Active Comparator): The instructor teaches the trainee in physical presence during the ERCP
  Interventions: Other: Training in presence of the instructor
- Telemedical training (Experimental): The instructor teaches the trainee telemedically by using smartglasses during the ERCP
  Interventions: Other: Telemedically training by an instructor

INTERVENTIONS:
Other: Training in presence of the instructor — The instructor gives the trainee instructions for the examination while he/she is present in the examination room.
  Arms: Training in presence
Other: Telemedically training by an instructor — The trainer gives instructions to the trainee through a telemedical connection to the examiner using SmartGlasses
  Arms: Telemedical training

SUMMARY:
The aim of this prospective randomized study is to evaluate whether telemedical assistance via SmartGlasses is equivalent to physical presence in teaching Endoscopic Retrograde Cholangiopancreaticography (ERCP) in terms of examination success and safety. Endoscopic papilla cannulation is a key skill for successful ERCP and therefore a measurable primary endpoint of the study. This can be measured as the time (in seconds/minutes) between stable visualization of the papilla and successful endoscopic cannulation of the target structure (bile duct or pancreatic duct).

DETAILED DESCRIPTION:
In sparsely populated regions of a country and where there is a lack of experienced specialists, it may not always be possible to have an experienced ERCP examiner present during an examination. Therefore, telemedical examination assistance via a connection to data glasses worn by the examiner is a possible option to replace the physical presence of an instructor or experienced ERCP examiner.

The aim of this prospective randomized study is to evaluate whether telemedical assistance via smart glasses is equivalent to physical presence in terms of examination success and safety. Endoscopic papilla cannulation is a key skill for successful ERCP and therefore a measurable primary endpoint of the study. This can be measured as the time (in seconds/minutes) between stable visualization of the papilla and successful endoscopic cannulation of the target structure (bile duct or pancreatic duct).

In addition to other efficacy endpoints, adverse events, which are expected to be rare, will be documented at 48-hour intervals and calculated as a rate. Telemedical 'live' support of an ERCP via data glasses has not yet been demonstrated or tested in a trial. To ensure the safety of the examination under these circumstances, the training examiner is present in the neighbouring room and can physically assist or take over the examination at any time if necessary.

ELIGIBILITY:
Inclusion criteria

* Adult patients aged ≥ 18 years without previous papillotomy Exclusion criteria
* Cannulation of the minor papilla necessary
* Significant comorbidity
* Haemodynamic instability
* Pregnant women
* Refusal or inability to give written informed consent for the study
* Instructor had to perform the examination himself/herself

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Papilla cannulation time | During the intervention: from the stable visualisation of the papilla until the successful cannulation of the papilla, assessed up to 60 minutes
  Time to cannulate the native papilla during ERCP

SECONDARY OUTCOMES:
Adverse events during and after ERCP | Time interval between insertion of the endoscope through the mouth up to 48 hours after ERCP
  All adverse events that occur during ERCP and after ERCP: number (n)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Schmitz, Dr.med., Principal Investigator — Helios Kliniken Schwerin
Locations (1):
- Helios Kliniken Schwerin, Schwerin, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: Yes
It is planned to share the IPD in a public repository such as re3data.org
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately after acceptance of the manuscript for publication
Access Criteria: No limitation

REFERENCES:
- [Background] Pan Y, Zhao L, Leung J, Zhang R, Luo H, Wang X, Liu Z, Wan B, Tao Q, Yao S, Hui N, Fan D, Wu K, Guo X. Appropriate time for selective biliary cannulation by trainees during ERCP--a randomized trial. Endoscopy. 2015 Aug;47(8):688-95. doi: 10.1055/s-0034-1391564. Epub 2015 Mar 6. PMID 25750038
- [Background] Testoni PA, Mariani A, Aabakken L, Arvanitakis M, Bories E, Costamagna G, Deviere J, Dinis-Ribeiro M, Dumonceau JM, Giovannini M, Gyokeres T, Hafner M, Halttunen J, Hassan C, Lopes L, Papanikolaou IS, Tham TC, Tringali A, van Hooft J, Williams EJ. Papillary cannulation and sphincterotomy techniques at ERCP: European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2016 Jul;48(7):657-83. doi: 10.1055/s-0042-108641. Epub 2016 Jun 14. PMID 27299638
- [Background] Biancheri P, Soriani P, Gabbani T, Bonura GF, Manno M. Smart glasses: Taking GI endoscopy to the metaverse era. Dig Liver Dis. 2023 May;55(5):692-693. doi: 10.1016/j.dld.2023.02.001. Epub 2023 Feb 26. No abstract available. PMID 36849287